CLINICAL TRIAL: NCT03603366
Title: Patient-centred Benefit-risk Observational Study of Low-dose Aspirin for CVD (Cardiovascular Disease) and CRC (Colorectal Cancer) Prevention
Brief Title: Study to Evaluate How Patients Regard the Benefits and Risks of Low-dose Aspirin for the Prevention of Heart and Blood Vessels Disease and for the Prevention of Cancer of the Colon and Rectum
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20211
Record Dates: First submitted 2018-07-20; First posted 2018-07-27 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Disease; Colorectal Cancer
MeSH Terms: conditions — Cardiovascular Diseases; Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary prevention: Patients in Italy who are eligible to use low-dose aspirin for primary prevention of CVD and CRC.
  Subgroups:
  * Patients eligible for and using low-dose aspirin who are at 20% ten-year CVD risk for primary prevention of CVD
  * Patients eligible for and not using low-dose aspirin who are at 20% ten-year CVD risk for primary prevention of CVD
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYE4465)
- Secondary prevention: Patients in Italy who are eligible to use low-dose aspirin for secondary prevention of CVD and CRC.
  Subgroups:
  * Patients eligible for and using low-dose aspirin for secondary prevention of CVD
  * Patients eligible for and not using low-dose aspirin for secondary prevention of CVD
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYE4465)
- Physicians: Physicians from Italy with experience recommending low-dose aspirin for primary and/or secondary prevention of CVD and CRC.

INTERVENTIONS:
Drug: Acetylsalicylic acid (Aspirin, BAYE4465) — This study does not involve prescription of the drugs. This study is a cross-sectional survey of patients taking low-dose aspirin or patients who are eligible but not taking low-dose aspirin.
  Other Names: Low-dose Aspirin
  Groups: Primary prevention; Secondary prevention

SUMMARY:
Research shows that low-dose Aspirin prevents diseases of heart and blood vessels as well as cancer of the colon and rectum and it is also associated with risk of bleeding. In this study, they want to learn how patients regard the benefits and risks of low-dose Aspirin for the prevention of these diseases. The researchers also want to learn how patients balance these risks and benefits.

ELIGIBILITY:
Patient Eligibility Criteria

Inclusion Criteria:

* Age and CVD characteristics

  * Primary prevention:

    * 50-70 years of age
    * Self-report clinical characteristics that result to 20% or higher, 10-year risk of CVD based on the Progetto Cuore scores
  * Secondary prevention:

    * 18 years or older
    * Having a self-reported history of CV event (e.g., myocardial infarction (MI), ischaemic stroke or Transient Ischaemic stroke, , and angina)
* Able to read and understand Italian
* No participation in an investigational program with interventions outside of routine clinical practice
* For qualitative interviews:

  * Willing and able to provide (electronic) informed consent to participate in the study
  * Willing and able to participate in a telephone interview, and to be audio-recorded
* For pilot/cognitive interviews :

  * Willing and able to complete an online survey
  * Willing and able to provide (electronic) informed consent to participate in the study
  * Willing and able to participate in an in-person interview, and to be audio-recorded
* For quantitative main survey:

  * Willing and able to complete an online survey
  * Willing and able to provide (electronic) informed consent to participate in the study

Exclusion Criteria:

* Have glucose-6-phosphate dehydrogenase (G6PD) deficiency (which commonly causes haemolytic anaemia, which is often triggered from eating fava beans, a condition called Favism)
* Have the following conditions (which are contraindications to low-dose aspirin)

  * Known hypersensitivity to salicylates
  * Known to have had asthma induced by salicylates
  * Having been diagnosed with acute gastroduodenal ulcers
  * Haemorrhagic diathesis
  * Renal failure
  * Hepatic failure
* Concomitant treatment with methotrexate
* Cognitive impairment, hearing difficulty, visual impairment, acute psychopathology, or insufficient knowledge of Italian that-in the opinion of the investigator/interviewer-could interfere with a patient's ability to provide written consent and complete an interview or survey
* To be currently pregnant
* Are pharmaceutical company employees or employed in a position where they have a direct role in treating patients with CVD

Physician Eligibility Criteria:

* A medically trained physician
* Able to read, speak, and understand Italian sufficiently to complete an interview
* Able to provide informed consent electronically
* Have at least five year experience prescribing low-dose aspirin for primary and secondary prevention of CVD
* Willing to be audio-recorded, including adherence to the interview instructions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are eligible for and/or taking low-dose aspirin will be recruited for qualitative interviews, pilot/cognitive interviews, and the main quantitative survey. Medically trained physicians who have experience prescribing low-dose aspirin for CVD (cardiovascular disease) and CRC (colorectal cancer) prevention will be eligible for the qualitative interviews.
Sampling Method: Non-Probability Sample
Enrollment: 1028 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Perceive of low dose aspirin | Up to 1 hour
  Using qualitative interviews to assess how patients and physicians perceive the benefits and risks of low-dose aspirin for the prevention of cardiovascular disease (CVD) and colorectal cancer (CRC)
Patients' benefit/risk trade-offs | Up to 1 hour
  Using quantitative surveys to elicit patients' benefit/risk trade-offs on key efficacy and safety outcomes of low-dose aspirin in CVD and CRC prevention

SECONDARY OUTCOMES:
Change in likelihood of AEs | Up to 1 hour
  Quantify the change in likelihood of adverse events (AEs) that patients are willing to accept in order to experience the benefits of low-dose aspirin for CRC and CVD prevention compared to CVD prevention alone
Preferences of aspirin using in different subgroups | Up to 1 hour
  Assess how different subgroups of patients, such as those using low-dose aspirin and those eligible for but not using low-dose aspirin, differ in their preferences

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/